CLINICAL TRIAL: NCT00918931
Title: Evaluation of Obatoclax Mesylate as Therapy for Patients With Systemic Mastocytosis
Brief Title: Obatoclax for Systemic Mastocytosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Gemin X (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0792
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Results first posted 2011-04-25 (Estimated); Last update posted 2011-11-04 (Estimated); Status verified 2011-10

CONDITIONS: Leukemia; Systemic Mastocytosis
Keywords: Leukemia; Systemic Mastocytosis; SM; Obatoclax mesylate; GX15-070MS
MeSH Terms: conditions — Leukemia; Mastocytosis, Systemic | interventions — obatoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Obatoclax Mesylate (Experimental): 30 mg by vein over 3 hours Days 1-3, 14-day cycle
  Interventions: Drug: Obatoclax Mesylate

INTERVENTIONS:
Drug: Obatoclax Mesylate — 30 mg given by vein over 3 hours on Days 1-3 of each 14-day study cycle.

SUMMARY:
The goal of this clinical research study is to learn if obatoclax mesylate can help to control systemic mastocytosis. The safety of this drug will also be tested.

DETAILED DESCRIPTION:
The Study Drug:

Obatoclax mesylate is designed to block the growth of malignant mast cells. This may cause cancer cells to die.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive obatoclax mesylate through a peripheral intravenous catheter (a needle in the vein of your arm). The drug will be given over 3 hours each day on Days 1-3 of each 14-day study cycle.

If the study doctor thinks it is needed, you might receive the study drug though a silicone-based central venous catheter (CVC). A central venous catheter is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. Some catheters cannot be used with the study drug. If you already have one of these catheters in your body, it may need to be replaced before you can begin receiving the study drug. You will sign a separate consent that will describe the procedure and its risks in detail.

Study Visits:

One (1) time during each study cycle, the following tests and procedures will be performed:

* You will be asked about any side effects you may be having and about any other drugs you may be taking.
* Blood (about 2 tablespoons) will be drawn for routine tests.

Every 3 months while you are taking the study drug, you will have a bone marrow biopsy/aspirate to check the status of the disease.

Length of Study:

You will be able to continue receiving the study drug for as long as you are benefitting. You will be taken off study if you have intolerable side effects or if the disease gets worse.

Follow-Up:

Three months after your last dose of study drug, your doctor will call you to ask you how you are feeling. This call should take about 10 minutes.

Additional Information:

* You must tell your doctor about any drug allergies you may have.
* You must tell your doctor about how much alcohol you consume and about any other drugs you may be taking, including vitamins, herbal remedies, and over-the-counter, prescription, and/or illegal drugs. Some of these will interact with the study drug.
* You must arrange to have someone drive you home after each treatment. You must not drive or operate machinery (including kitchen appliances) after you have received the study drug until any possible side effects have gone away.
* If you feel you any side effects or symptoms while you are on study, you must contact your doctor right away.

This is an investigational study. Obatoclax mesylate is not FDA approved or commercially available. At this time, obatoclax mesylate is only being used in research.

Up to 25 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Systemic Mastocytosis (SM); including mast cell leukemia.
2. Age equal to or greater than 18 years
3. Minimum of two weeks since any major surgery or completion of radiation
4. Eastern Cooperative Oncology Group (ECOG) performance status equal to or less than 2
5. Adequate liver function as shown by serum bilirubin equal to or less than 1.5 * upper limit of normal (ULN), and serum alanine aminotransferase (ALT) equal to or less than 3 * ULN.
6. Signed informed consent

Exclusion Criteria:

1. Patients with low blood cell counts (Grade 3 or 4), unless it is known that the low blood cell count is due to systemic mastocytosis.
2. Treatment with any conventional (specifically, interferon or cladribine) or investigational medicine for SM within the preceding 4 weeks
3. Chronic treatment with systemic steroids (unless limited to 10 mg prednisone equivalent per day or less) or another immunosuppressive agent
4. Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin. Patient may have SM-associated clonal hematologic disease that does not require therapy, as judged by the treating physician and approved by the principal investigator).
5. Other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study as judged by the Principal Investigator (i.e., severely impaired lung function, uncontrolled diabetes, uncontrolled hypertension, severe infection, severe malnutrition, unstable angina, or congestive heart failure - New York Heart Association Class III or IV, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within six months, chronic liver or renal disease, active upper GI tract ulceration)
6. A known history of human immunodeficiency virus (HIV) seropositivity
7. Women who are pregnant or breast feeding,or women/men able to conceive and unwilling to practice an effective method of birth control. Women of childbearing potential must have a negative urine or serum pregnancy test within 48 hours prior to administration of obatoclax. Women of childbearing potential is defined as women who have not undergone a hysterectomy or bilateral oophorectomy, has not been naturally postmenopausal for at least 24 consecutive months.
8. Patients with a known hypersensitivity to obatoclax mesylate or to its excipients (PEG 300 and Tween 20)
9. Patients unwilling to or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srdan Verstovsek, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 6/5/2009 through 3/18/2010. All participants recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Three patients were registered and all of them received treatment.
Period: Overall Study
Arm/Group | Obatoclax Mesylate
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Obatoclax Mesylate
Number analyzed (Participants) | 3
Age Continuous [Median (Full Range); unit: years] | 75 [60 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Response rate is defined as number of participants with objective response divided by number of participants evaluated. Objective response is complete response and partial response where 'complete response' constitutes total elimination of a symptom or sign of the disease; 'partial response' constitutes at least 50% improvement in a symptom or sign of the disease. Objective response definitions of response evaluated following guidelines proposed by Valent et al. (International working group consensus criteria).
Time Frame: 3-Month Response Evaluation
Population: Analysis was per protocol.
Measure: Number; unit: participants
Arm/Group | Obatoclax Mesylate
Number analyzed (Participants) | 3
participants | 0

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Obatoclax Mesylate
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obatoclax Mesylate (N=3)
Anorexia (Gastrointestinal disorders) | 2 (2)
Ataxia (Nervous system disorders) | 1 (3)
Confusion (Nervous system disorders) | 1 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 2 (5)
Injection site reaction (General disorders) | 1 (1)
Memory Impairment (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (4)
Puritis (Skin and subcutaneous tissue disorders) | 1 (1)
Psychosis (Nervous system disorders) | 1 (2)
Mood Alteration (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes